CLINICAL TRIAL: NCT00096629
Title: Injection of Renal Cell Carcinoma Patients With Human and Mouse Prostate Specific Membrane Antigen (PSMA) DNA: A Phase I Trial to Assess Safety and Immune Response
Brief Title: Vaccine Therapy in Treating Patients With Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 03-125; MSKCC-03125
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

ARMS (2):
- human PSMA (Experimental): Patients will receive a total of 6 vaccinations via the intramuscular route. Sites of injection should have intact lymphatic drainage. Groups of six patients will be randomized at each dose level, 3 for each arm, to receive either three immunizations with mouse PSMA followed by three immunizations with human PSMA or three immunizations with human PSMA followed by three immunizations with mouse PSMA.
  Interventions: Biological: human prostate-specific membrane antigen plasmid DNA vaccine; Biological: mouse prostate-specific membrane antigen plasmid DNA vaccine
- mouse PSMA (Experimental): Patients will receive a total of 6 vaccinations via the intramuscular route. Sites of injection should have intact lymphatic drainage. Groups of six patients will be randomized at each dose level, 3 for each arm, to receive either three immunizations with mouse PSMA followed by three immunizations with human PSMA or three immunizations with human PSMA followed by three immunizations with mouse PSMA.
  Interventions: Biological: human prostate-specific membrane antigen plasmid DNA vaccine; Biological: mouse prostate-specific membrane antigen plasmid DNA vaccine

INTERVENTIONS:
Biological: human prostate-specific membrane antigen plasmid DNA vaccine
Biological: mouse prostate-specific membrane antigen plasmid DNA vaccine

SUMMARY:
RATIONALE: Vaccines made from DNA may make the body build an immune response to kill tumor cells.

PURPOSE: This randomized phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of vaccination with human and mouse prostate-specific membrane antigen (PSMA) DNA in patients with renal cell carcinoma.
* Determine the maximum tolerated dose of this regimen in these patients.
* Determine antibody responses to human PSMA in patients treated with this regimen.

Secondary

* Assess antitumor response in patients treated with this regimen.

OUTLINE: This is a randomized, dose-escalation study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive human prostate-specific membrane antigen (PSMA) DNA vaccine intramuscularly (IM) once every 3 weeks for 3 doses (doses 1-3). Patients then receive mouse PSMA DNA vaccine IM once every 3 weeks for 3 doses (doses 4-6).
* Arm II: Patients receive mouse PSMA DNA vaccine IM once every 3 weeks for 3 doses (doses 1-3). Patients then receive human PSMA DNA vaccine IM once every 3 weeks for 3 doses (doses 4-6).

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive additional booster vaccinations with the second form of PSMA DNA vaccine received (for doses 4-6) every 8 weeks for up to 4 additional doses.

Cohorts of 3-6 patients per arm receive escalating doses of human and mouse PSMA DNA vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma
* Patients with minimal disease burden are eligible provided they meet one or more of the following criteria:

  * Prior nephrectomy and completely resected metastases
  * Favorable-risk group, as defined by all of the following criteria:

    * Karnofsky 80-100%
    * Hemoglobin ≥ 13 g/dL (male) or ≥ 12 g/dL (female)
    * Corrected calcium ≤ 10 mg/dL
    * Prior nephrectomy
    * Serum lactate dehydrogenase ≤ 200 μ/L
  * Prior nephrectomy with metastases confined to lung and/or small volume metastatic disease (< 3 cm) exclusive of bone and liver
* No spinal, epidural, or CNS lesions
* No bone, liver or brain disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* See Disease Characteristics
* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* WBC ≥ 3,500/mm^3
* Hemoglobin ≥ 12.0 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 2.0 mg/dL
* SGOT < 3.0 times upper limit of normal

Renal

* See Disease Characteristics
* Creatinine ≤ 2.0 mg/dL OR
* Creatinine clearance ≥ 40 mL/min

Cardiovascular

* No clinically significant cardiac disease
* No New York Heart Association class III or IV heart disease

Pulmonary

* No severe debilitating pulmonary disease

Other

* Fertile patients must use effective contraception
* No other active secondary malignancy within the past 5 years except non-melanoma skin cancer
* No infection requiring antibiotic treatment
* No narcotic- or steroid-dependent pain

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy

Endocrine therapy

* At least 4 weeks since prior corticosteroid therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy to only measurable lesion

Surgery

* See Disease Characteristics
* No concurrent surgery

Other

* Recovered from all prior therapy
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
safety | 2 years
feasibility | 2 years

SECONDARY OUTCOMES:
antibody responses | 2 years
anti-tumor response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slovin, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/